CLINICAL TRIAL: NCT01203943
Title: A Phase 2 Sequential, Ascending Dose Study to Characterize the Safety, Tolerability, Pharmacokinetic and Biological Activity of CC-930 in Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Study to Characterize the Safety, PK and Biological Activity of CC-930 in Idiopathic Pulmonary Fibrosis (IPF)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The benefit/ risk profile does not support continuation of this study.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-930-IPF-001
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Fibrosis; Interstitial Lung Disease; Lung Diseases, Interstitial
Keywords: Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Fibrosis; Interstitial Lung Disease; Lung Diseases, Interstitial; CC-930
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Fibrosis; Lung Diseases, Interstitial | interventions — 4-(9-(tetrahydrofuran-3-yl))-8-(2,4,6-trifluorophenylamino)-9H-purin-2-ylaminocyclohexan-1-ol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): • Cohort 1: CC-930 50 mg PO daily (two 25 mg capsules once per day PO) beginning on Day 1 in the AM.
  Interventions: Drug: CC-930
- Cohort 2 (Experimental): • Cohort 2: CC-930 100 mg PO daily (one 100 mg capsule once per day PO) beginning on Day 1 in the AM
  Interventions: Drug: CC-930
- Cohort 3 (Experimental): • Cohort 3: CC-930 100 mg twice daily approximately 12 hours apart (one 100 mg capsule twice per day PO) beginning on Day 1.
  Interventions: Drug: CC-930
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CC-930 — CC-930 50 mg PO daily up to 56 weeks beginning on Day 1
  Arms: Cohort 1
Other: Placebo — Placebo
  Arms: Placebo
Drug: CC-930 — CC-930 100 mg PO daily up to 56 weeks beginning on Day 1
  Arms: Cohort 2
Drug: CC-930 — C-930 100 mg twice daily approximately 12 hours apart up to 56 weeks beginning on Day 1
  Arms: Cohort 3

SUMMARY:
The primary purpose of the study is to evaluate the safety and PK profile of CC-930 in idiopathic pulmonary fibrosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of non-childbearing potential ≥50 years of age (at the time of signing the informed consent document) with documented IPF
* Diagnosis of IPF based on current ATS/ERS guidelines

  * Usual interstitial pneumonia (UIP) pattern on HRCT and/or UIP pattern on histopathology (ie surgical lung biopsy), and
  * Exclusion of known causes of interstitial lung disease (such as environmental exposure, connective tissue disease and drug toxicity), Or
  * UIP pattern on surgical lung biopsy required if HRCT is inconsistent with UIP

Exclusion Criteria:

* FVC : < 50% predicted >90% predicted
* DLco:< 25% predicted >90% predicted
* Saturated oxygen (SpO2) of <92% (room air [sea level] at rest). SpO2 of < 88% (room air [≥ 5,000 feet above sea level (1524 meters]) at rest)
* Use of any cytotoxic/immunosuppressive agent (other than prednisone ≤ 12.5 mg/day or equivalent) including, but not limited to, azathioprine, cyclophosphamide, methotrexate and cyclosporine within 4 weeks of screening
* Use of any cytokine modulators:

  * Use of any biologic agent (such as etanercept, adalimumab, efalizumab, infliximab, golimumab, certolizumab) within 12 weeks or five half-lives of screening, and in the case of rituximab, use within 24 weeks of screening or no recovery of CD 19-positive B lymphocytes if the last dose of rituximab has been more than 24 weeks prior to screening
  * Alefacept within 24 months of randomization
* Use of any therapy targeted to treat IPF (including but not limited to d-penicillamine, endothelium receptor antagonist [eg bosentan, ambrisentan], interferon gamma-1B, pirfenidone) within 4 weeks of screening
* Use of n-acetylcysteine (NAC) for IPF (≥1800 mg/day) within 4 weeks of screening
* Use of any investigational drug within one month of screening, or 5 PD/PK half lives, if known (whichever is longer)
* Current smoker

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2012-01-31 (Actual); Study Completion 2012-08-24 (Actual)

PRIMARY OUTCOMES:
Safety | Week 4
  Number of participants with adverse events

SECONDARY OUTCOMES:
Long-term safety | Weeks 52-104
  Number of participants with adverse events
Disease progression/death rates | Up to week 56
  Time to disease progression and death
Disease progression/death rates | Weeks 52-104
  Time to disease progression and death from week 52
Pharmacokinetics-Cmax | Week 1 (baseline) and week 2
  Maximum observed concentration in plasma
Pharmacokinetics-Cmin | Week 0 (baseline) and week 2
  Minimum observed concentration in plasma
Pharmacokinetics-AUC | Week 0 (baseline) and week 2
  Area under the plasma concentration - time curve
Pharmacokinetics-Tmax | Week 0 (baseline) and week 2
  Time to reach Cmax
Pharmacokinetics - t 1/2 | Week 0 (baseline) and week 2
  Terminal half-life (t1/2)
Pharmacokinetics-Vz/f | Week 0 (baseline) and week 2
  Apparent volume of distribution
Pharmacokinetics-CL/F | Week 0 (baseline) and week 2
  Apparent total body clearance

CONTACTS AND LOCATIONS:
Overall Officials: William Smith, MD, Study Director — Celgene Corporation
Locations (22):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC Davis Medical Center, Division of Pulmonary and Critical Care Medicine, Sacramento, California
  - Stanford University, Pulmonary & Critical Care Clinic, Stanford, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Louisville, Louisville, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Geisenger Center for Clinical Studies, Danville, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Vermont Lung Center, Colchester, Vermont
- Canada (6):
  - University of Calgary, Peter Lougheed Centre, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital/University of British Columbia, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Victoria Hospital, London, Ontario
  - Notre-Dame Hospital du CHUM, Montreal, Quebec

REFERENCES:
- [Background] van der Velden JL, Ye Y, Nolin JD, Hoffman SM, Chapman DG, Lahue KG, Abdalla S, Chen P, Liu Y, Bennett B, Khalil N, Sutherland D, Smith W, Horan G, Assaf M, Horowitz Z, Chopra R, Stevens RM, Palmisano M, Janssen-Heininger YM, Schafer PH. JNK inhibition reduces lung remodeling and pulmonary fibrotic systemic markers. Clin Transl Med. 2016 Dec;5(1):36. doi: 10.1186/s40169-016-0117-2. Epub 2016 Sep 2. PMID 27590145